CLINICAL TRIAL: NCT03667339
Title: Direct Anterior Total Hip Arthroplasty (THA), in Versus Outpatients : A Prospective Monocentric Study in Rennes University Hospital.
Acronym: AHVACA
Status: Terminated | Type: Observational
Why Stopped: lack of recruitment
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3084_AHVACA
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Direct Anterior Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- outpatients group: Patient schedulded to undergo outpatient Direct Anterior Total Hip Arthroplasty
  Interventions: Procedure: Direct Anterior Total Hip Arthroplasty
- inpatients group: Patient schedulded to undergo inpatient Direct Anterior Total Hip Arthroplasty
  Interventions: Procedure: Direct Anterior Total Hip Arthroplasty

INTERVENTIONS:
Procedure: Direct Anterior Total Hip Arthroplasty — Direct Anterior Total Hip Arthroplasty

SUMMARY:
The main objective is to show that cumulative length of stay over the first 45 post operative days (i.e. : primary length of stay and readmission) is significantly lower in the outpatients group than in the inpatients group

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary total hip arthroplasty for hip osteoarthritis, primary or secondary osteoarthritis (dysplasia or post-traumatic) or osteonecrosis
* Good enough understanding of outpatient management and patient adherence to post-operative instructions
* Sufficient patient complicance to medical orders
* Living and hygiene conditions, at least, equivalent to the ones the hospital provides
* To be of age
* Non opposition to the protocole participation

Outpatients group :

- Patient schedulded to undergo outpatient THA

Inpatients group :

- Patient schedulded to undergo inpatient THA because of not fiting the following items :

* Less than an hour distance of a Health Center that provides appropriate care with regard to the surgery
* Rapid access to a phone
* Designated driver and caretaker available (at least the first night after discharge from the hospital) after the procedure Or turning down outpatient THA

Exclusion Criteria:

* Anaesthetic point of view :

  * ASA physical status ≥ 3 and : unstabilize disease with appropriate treatment or lack of preoperative mutual agreement between anesthesiologist and surgeon or not inconsiderable interaction between the operation and the disease or its treatment
  * Pre-operative Hb < 12 (♀) < 13 (♂) g/L (NB : no Hb control before discharge except if excessive blood loss ; Hb < 10g/L contraindicates outpatient surgery)
  * Opioid chronic pre-operative therapy or opioid addiction
* Surgical point of view :

  * Ambulatory pre-operative status requiring use of two crutches or walking frame / distance walked < 30 m
  * THA procedure for femoral neck fracture requiring
  * Additional operative technic needed
* Adult safeguarding.

Exclusion criteria applies to all in and outpatients.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with Direct Anterior Total Hip Arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Cumulative lenght of stay | 45 days before surgery
  Cumulative lenght of stay ( ie : the sum of the days of hospitalization corresponding to the initial hospitalization and readmissions if there are any)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis POLARD, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France